CLINICAL TRIAL: NCT00969189
Title: A Cohort Evaluation of the Pediatric Igel Airway in 200 Children and in 50 Infants
Brief Title: Evaluation of the Pediatric Igel Airway in 250 Children
Status: Terminated | Type: Observational
Why Stopped: Initial number of 250 was not based on sample size. Most airway studies use n=100 therefore trial stopped when 120 children recruited
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Royal United Hospital Bath NHS Trust (Other)
Responsible Party: Principal Investigator, Michelle White, Consultant in Paediatric Anaesthesia and Critical Care, University Hospitals Bristol and Weston NHS Foundation Trust
Other Study IDs: CH/2008/2808; NRES ID: 08/H0101/198
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Anesthesia; Child; Infant
Keywords: anesthesia; child; infant; laryngeal mask

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children: between 10 and 30 kgs
- Infants: between 5 - 10 kg

SUMMARY:
Once a child has been anaesthetised and is fully asleep, a special airway tube called a laryngeal mask is often inserted into their mouth to help with their breathing. This tube is removed just before the child wakes up.

A new type of airway tube, called an i-gel airway, has been developed for children, which is hoped will be easier to insert, safer once in position, and will be less likely to cause a sore throat after the anaesthetic than a standard laryngeal mask. The adult i-gel airway has been available for adults since 2007, and early trials have shown very encouraging results.

ELIGIBILITY:
Inclusion Criteria:

* All children weighing 5 -30kg
* Classified by the American Society of Anesthesiology (ASA) as grade 1-2,
* Scheduled for elective surgery under general anaesthesia, in whom a LMA or PLMA would otherwise be used for airway maintenance and in whom neuromuscular blocking drugs will not be used.

Exclusion Criteria:

* Inability of patient or parents to understand the study or consent process
* Neck pathology
* Previous or anticipated airway problems
* Pathology of airway, respiratory tract, upper gastrointestinal tract
* Increased risk of regurgitation or aspiration
* Weight >30kg or <5 kg
* ASA 3 and above,
* Emergency surgery

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children between 10 - 30 kgs infants between 5-10 kgs
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Does the i-gel (a new supraglottic airway device) perform adequately in anaesthetised healthy children? | during anaesthesia

SECONDARY OUTCOMES:
Ease of insertion, Complication rates and manipulation rates during use, Airway seal pressure, Effective ventilation, Post-operative sequelae | during anaesthesia and up to 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michelle White, MB ChB, Principal Investigator — UH Bristol NHS Foundation Trust
Locations (1):
- UH Bristol NHS Foundation Trust, Bristol, Avon, United Kingdom